CLINICAL TRIAL: NCT00900445
Title: Impact of Obesity on the Pharmacokinetics of Anticancer Therapy in Children With High Risk Acute Lymphoblastic Leukemia (ALL)
Brief Title: Studying Body Mass Index in Younger Patients Who Are Receiving Treatment for High-Risk Acute Lymphoblastic Leukemia
Status: Withdrawn | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACCL0631; NCI-2011-02151 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000588173; ACCL0631 (Other: Childrens Oncology Group); COG-ACCL0631 (Other: DCP); ACCL0631 (Other: CTEP); U10CA095861 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2013-03

CONDITIONS: Acute Lymphoblastic Leukemia; Untreated Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Daunorubicin; Prednisolone; Methylprednisolone; Prednisone; deltacortene; prednylidene; Vincristine

GROUPS / COHORTS (1):
- Basic science (pharmacokinetics): Patients receive anticancer therapy as prescribed by their treating clinicians. Patients receive prednisone/prednisolone orally twice on either day 1 or day 8. Patients also receive daunorubicin hydrochloride IV over 30 minutes and vincristine IV once on the same day.
  Interventions: Drug: Daunorubicin Hydrochloride; Other: Pharmacological Study; Drug: Prednisolone; Drug: Prednisone; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Other: Pharmacological Study — Correlative studies
Drug: Prednisolone — Given orally
  Other Names: (11beta)-11,17,21-Trihydroxypregna-1,4-diene-3,20-dione; .delta.1-Hydrocortisone; Adnisolone; Aprednislon; Capsoid; Cortalone; Cortisolone; Dacortin H; Decaprednil; Decortin H; Delta(1)Hydrocortisone; Delta- Cortef; Delta-Cortef; Delta-Diona; Delta-F; Delta-Phoricol; Delta1-dehydro-hydrocortisone; Deltacortril; Deltahydrocortisone; Deltasolone; Deltidrosol; Dhasolone; Di-Adreson-F; Dontisolon D; Estilsona; Fisopred; Frisolona; Gupisone; Hostacortin H; Hydeltra; Hydeltrasol; Klismacort; Kuhlprednon; Lenisolone; Lepi-Cortinolo; Linola-H N; Linola-H-Fett N; Longiprednil; Metacortandralone; Meti Derm; Meticortelone; Opredsone; Panafcortelone; Precortisyl; Pred-Clysma; Predeltilone; Predni-Coelin; Predni-Helvacort; Prednicortelone; Prednisolonum; Prelone; Prenilone; Sterane
Drug: Prednisone — Given orally
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This clinical trial is studying body mass index in younger patients receiving prednisone/prednisolone, vincristine, daunorubicin, and pegaspargase for high-risk acute lymphoblastic leukemia. Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about the affect of body mass index on the way anticancer drugs work in the body. It may also help doctors predict how patients will respond to treatment

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the pharmacokinetics of prednisone/prednisolone, vincristine, and daunorubicin hydrochloride among obese, middle-weight, and underweight children aged 10 to less than 20 years of age undergoing induction therapy for high-risk acute lymphoblastic leukemia.

II. To examine the relationship between the above parameters and response status as defined by early response and induction failure

OUTLINE: This is a multicenter study. Patients are stratified according to body mass index (BMI) (greater than or equal to 95th percentile [obese] vs 10th to 95th percentile [normal or at risk for overweight] vs less than or equal to 10th percentile [underweight]).

Patients receive anticancer therapy as prescribed by their treating clinicians. Patients receive prednisone/prednisolone orally twice on either day 1 or day 8. Patients also receive daunorubicin hydrochloride IV over 30 minutes and vincristine IV once on the same day.

Blood samples are obtained on either day 1 or day 8** of induction therapy for pharmacokinetic analysis of prednisone, daunorubicin hydrochloride, and vincristine activity levels.

Blood samples are analyzed via high-performance liquid chromatography (HPLC), ultrafiltration, a Nessler reaction, ELISA, and liquid chromatography using reverse-phase chromatography, fluorescent detection, and solid-phase extraction.

Demographic information, including ethnicity, is also collected. Weight and height is recorded at diagnosis and on the day pharmacokinetic assessment of vincristine, prednisone, and daunorubicin hydrochloride begins.

NOTE: **Patients who are being sampled on day 8 of induction therapy and who have received intravenous corticosteroid therapy in the first week of induction must have received at least six oral prednisone/prednisolone doses prior to the morning prednisone/prednisolone dose on day 8.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be newly diagnosed with acute lymphoblastic leukemia and the intended induction treatment must contain prednisone/prednisolone, vincristine and daunorubicin in the doses and schedule as per the current COG AALL0232 protocol; prior registration onto a COG protocol is not required
* Patients must be able to take either prednisone/prednisolone reliably by mouth on day 1 or 8 of induction (depending on sampling schedule chosen); patients who are being sampled on Induction day 8 and who have received intravenous corticosteroid therapy in the first week of induction must have received a minimum of six oral prednisone/prednisolone doses prior to the morning prednisone/prednisolone dose on induction day 8

Exclusion Criteria:

* Serum transaminase concentrations >= 5 X ULN for age
* Total serum bilirubin (conjugated + unconjugated) >= 1.5 mg/dl (>= 26 micromol/L)
* Serum creatinine > 1.5 X ULN for age
* With the exception of prednisone/prednisolone, receipt of medications or food known or with the potential to alter the pharmacokinetics of the drugs under study within 14 days of diagnosis and throughout the period of pharmacokinetic sampling; such agents include but are not limited to: grapefruit, tangelos or the juice of these fruits; St. Johns wort; anticonvulsants: carbamazepine, oxcarbazepine, phenytoin, phenobarbital, primidone; azole antifungal agents: ketoconazole, fluconazole, itraconazole, voriconazole; macrolide antibiotics: erythromycin, clarithromycin; isoniazid; rifampin; verapamil; and diltiazem
* Presence of known malabsorption syndrome
* Females with known pregnancy (pregnancy test must be negative to be eligible)

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-03-24 (Actual); Primary Completion 2009-08-17 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of prednisone/prednisolone | Pre-dose, 0.5, 1, 1.5, 2, 4, 6 to 8, 10 and 12 hours
  Two multiple comparisons (normal weight versus obese and normal weight versus underweight groups) will be conducted with a priori planned contrasts using the Bonferroni adjustment method.
Pharmacokinetic parameters of daunorubicin hydrochloride | Pre-dose, 0.5, 0.75, 1, 2, 4, 8, 12, 24 to 36 hours, and 48 to 72 hours
  Two multiple comparisons (normal weight versus obese and normal weight versus underweight groups) will be conducted with a priori planned contrasts using the Bonferroni adjustment method.
Pharmacokinetic parameters of vincristine sulfate | Pre-dose, 0.5, 1, 2, 4, 8, 24 to 36 hours, and 48 to 72 hours
  Two multiple comparisons (normal weight versus obese and normal weight versus underweight groups) will be conducted with a priori planned contrasts using the Bonferroni adjustment method.

SECONDARY OUTCOMES:
RER and SER status | Up to 1.5 years
  To examine the relationship between pharmacokinetic parameters and RER versus SER status, univariate and multiple logistic regressions will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Pollack, Principal Investigator — Children's Oncology Group
Locations (1):
- Childrens Oncology Group, Philadelphia, Pennsylvania, United States